CLINICAL TRIAL: NCT03156088
Title: Clinical and Urodynamic Predictors for Sacral Neuromodulation Outcomes in Patients With Overactive Bladder: A Cohort Study
Brief Title: Clinical and Urodynamic Predictors for Sacral Neuromodulation Outcomes in Overactive Bladder
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Amr AbdAllah AbdelMaboud Mohamed Mahran, Assistant lecturer of Urology, Assiut University
Other Study IDs: IRB000087517
Record Dates: First submitted 2017-05-13; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Overactive Bladder
Keywords: Predictors; Sacral neuromodulation; Outcomes; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Overactive Bladder Patients: Overactive bladder patients treated with sacral neuromodulator "InterStim"
  Interventions: Device: Sacral Neuromodulator "InterStim"

INTERVENTIONS:
Device: Sacral Neuromodulator "InterStim"

SUMMARY:
Overactive bladder syndrome (OAB) is a prevalent disorder that affects about 10% of the adult population and > 40% of elderly. It is defined by the presence of urgency, with or without urge incontinence, in the absence of infection or other pathology. In 1997 through 1999, sacral nerve stimulation SNS (InterStim, Medtronic Inc., Minneapolis, Minnesota) was approved by the U.S. Food and Drug Administration (FDA) for treating urge urinary incontinence, urinary urgency, and frequency. Despite the large numbers of SNS performed, the only objective clinical evaluation of OAB is urodynamic detrusor instability (UDI) with some evidence suggesting a correlation with outcomes after sacral neuromodulation.

Interestingly, the mechanism of action of SNS is not fully understood. Theories include direct activation of efferent fibers to the striated urethral sphincter causing reflex relaxation of the detrusor or potential activation of afferent fibers selectively which can lead to inhibition at spinal and supraspinal levels. Somatic sacral afferent inflow activation at sacral level affects the storage and emptying reflexes in the bladder and central nervous system, explaining the beneficial effects of neuromodulation on both storage and emptying functions of the bladder. Malaguti and his colleagues detected somatosensory evoked potentials during sacral neuromodulation, revealing that sacral neuromodulation works by both sacral afferent activity and somatosensory cortex activation. As sacral neuromodulation is clinically proven for both storage and emptying bladder dysfunctions, it is difficult to isolate its action to either sacral afferent or efferent circuits in the micturition reflex pathway. In our study, we are going to study sacral neuromodulation outcome predictors from the clinical and urodynamic perspectives in order to help identifying the right candidates for sacral neuromodulation procedure.

DETAILED DESCRIPTION:
1.0 Introduction: Overactive bladder syndrome (OAB) is a prevalent disorder that affects about 10% of the adult population and > 40% of elderly. It is defined by the presence of urgency, with or without urge incontinence, in the absence of infection or other pathology. In 1997 through 1999, sacral nerve stimulation SNS (InterStim, Medtronic Inc., Minneapolis, Minnesota) was approved by the U.S. Food and Drug Administration (FDA) for treating urge urinary incontinence, urinary urgency, and frequency. Despite the large numbers of SNS performed, the only objective clinical evaluation of OAB is urodynamic detrusor instability (UDI) with some evidence suggesting a correlation with outcomes after sacral neuromodulation.

Interestingly, the mechanism of action of SNS is not fully understood. Theories include direct activation of efferent fibers to the striated urethral sphincter causing reflex relaxation of the detrusor or potential activation of afferent fibers selectively which can lead to inhibition at spinal and supraspinal levels. Somatic sacral afferent inflow activation at sacral level affects the storage and emptying reflexes in the bladder and central nervous system, explaining the beneficial effects of neuromodulation on both storage and emptying functions of the bladder. Malaguti and his colleagues detected somatosensory evoked potentials during sacral neuromodulation, revealing that sacral neuromodulation works by both sacral afferent activity and somatosensory cortex activation. As sacral neuromodulation is clinically proven for both storage and emptying bladder dysfunctions, it is difficult to isolate its action to either sacral afferent or efferent circuits in the micturition reflex pathway. In our study, we are going to study sacral neuromodulation outcome predictors from the clinical and urodynamic perspectives in order to help identifying the right candidates for sacral neuromodulation procedure.

2.0 Specific Aims:

* Specific aim#1: Using the medical reporting systems, we will identify all patients who, underwent sacral neuromodulation at University Hospitals of Cleveland from January 1, 2012 through February, 2017.
* Specific aim#2: Reporting on the efficacy outcomes including: rate of successful placement, rate of reported patient improvement after peripheral nerve (PNE) stage 1 and stage 2 procedure. The proportion of patients who undergo stage 2 compared to patients who had PNE. Rate of removal after full implantation and rate of battery change. Finally, will report on patient satisfaction, change in disease-specific severity scores and change in health-related quality of life
* Specific aim #3: Will identify preoperative clinical and urodynamic factors that can predict successful outcome and or/ failure.
* Specific aim #4: to identify predictors in subgroups of patients with OAB including:

  1. Wet versus dry subgroups.
  2. With urodynamic detrusor instability (UDI) versus no UDI subgroups.
  3. Neurogenic versus non-neurogenic.
  4. Staged versus non-staged procedure.
* Specific aim #5: Validating the identified predictors in a different established set of patients from Cleveland Clinic.
* Specific aim#6: Reporting on safety outcomes including intraoperative complications, early postoperative complications (within 30 days) and later postoperative complications. A modified Dindo classification will be utilized.

3.0 Data management and analysis: Data collection: Data will be collected from the medical reporting systems (Ambulatory medical reporting system and physician portal), University Hospitals Cleveland Medical Center and affiliated Hospitals, Cleveland, OH.

Data storage: REDCap software will be used for data storage. Computer software: SPSS 24 will be used for statistical analysis. Statistical tests: Continuous characteristics will be summarized with mean, median, and range; categorical characteristics will be summarized with number and percentage. For specific aim#2 and #3, #4, #5: associations of baseline characteristics with outcomes will be further evaluated using univariate, and multivariate logistic regression models and summarized with odds ratios (ORs) and 95% confidence intervals (CIs). Model calibration will be evaluated using the Hosmer and Lemeshow goodness-of-fit test to identify the best model. The comparison will be performed using independent sample T -test for normally disturbed continuous variables and Wilcoxon test for skewed data. Chi-square tests will be used for comparing categorical variables. For specific aim#6, Cox proportional hazard models will be used to evaluate the predictors of failure after device implantation, we will be using Hosmer and Lemeshow goodness-of-fit test. All tests will be 2 sided; P values less than .05 were considered statistically significant. Statistical analyses will be performed using SAS software (SAS Institute, Inc, Cary, North Carolina).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult female at least 18 years old.
* Persistent symptoms in spite of the use of at least two anticholinergics
* Urodynamic assessment within the previous year prior to the procedure.

Exclusion Criteria:

* PVR >150 ml on 2 occasions within 6 months prior to the procedure.
* Surgically altered detrusor muscle, such as augmentation cystoplasty.
* Serum creatinine level greater than twice the upper limit of normal within the previous year prior to the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Under an approved institutional review board #01-16-48, the medical and surgical database will be used to identify all patients who had test stimulation, stage I and stage II sacral neuromodulation at University Hospitals, Cleveland between January 1 2012 through February 2017. The study protocol is designed in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Successful treatment | 12 months
  will be denoted by patient symptoms improvement and stage II InterStim. > 50 improvement of patient symptoms will be considered.
Treatment failure | 12 months
  if the patient has persistence of his/her symptoms, mild improvement, operation site pain or any other causes- which lead to device removal.

SECONDARY OUTCOMES:
Postoperative complications | Early < month and late > 1 month and up to 12 months
  Clavien-Dindo classification
SNM efficacy in those with prior Botox bladder injection | 12 months
  Success vs failure
Trends of failure and success in neurogenic versus non-neurogenic overactive bladder | 12 months
  Incidence
Trends of failure and success in in wet versus dry patients | 12 months
  Incidence
Trends of failure and success in staged versus non-staged procedure | 12 months
  Incidence "Change"
Incidence and predictors of reoperation after SNM | 12 months
  Incidence and prediction

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Result] Chapple CR, Artibani W, Cardozo LD, Castro-Diaz D, Craggs M, Haab F, Khullar V, Versi E. The role of urinary urgency and its measurement in the overactive bladder symptom syndrome: current concepts and future prospects. BJU Int. 2005 Feb;95(3):335-40. doi: 10.1111/j.1464-410X.2005.05294.x. PMID 15679789
- [Result] Hashim H, Abrams P. Is the bladder a reliable witness for predicting detrusor overactivity? J Urol. 2006 Jan;175(1):191-4; discussion 194-5. doi: 10.1016/S0022-5347(05)00067-4. PMID 16406907
- [Result] Malaguti S, Spinelli M, Giardiello G, Lazzeri M, Van Den Hombergh U. Neurophysiological evidence may predict the outcome of sacral neuromodulation. J Urol. 2003 Dec;170(6 Pt 1):2323-6. doi: 10.1097/01.ju.0000095921.81600.4d. PMID 14634406
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Result] Leng WW, Chancellor MB. How sacral nerve stimulation neuromodulation works. Urol Clin North Am. 2005 Feb;32(1):11-8. doi: 10.1016/j.ucl.2004.09.004. PMID 15698871
- See also: Accessed November, 11th 2015 — https://professional.medtronic.com/pt/uro/snm/edu/about/index.htm#.VkJ5NberTIU